CLINICAL TRIAL: NCT02110095
Title: Picosure Alexandrite Laser for the Treatment of Unwanted Tattoos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN14-PICO-MULTI-JD
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Results first posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-11

CONDITIONS: Unwanted Tattoos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Picosure Laser System (Experimental): Picosure Laser System for the treatment of unwanted tattoos
  Interventions: Device: Picosure Laser System

INTERVENTIONS:
Device: Picosure Laser System — Picosure Laser System for the Treatment of Unwanted Tattoos

SUMMARY:
The purpose of this study is to evaluate the Picosure Laser System for the treatment of unwanted tattoos.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or female between 18 and 85 years old.
2. Is willing to consent to participate in the study.
3. Is willing to comply with all requirements of the study including being photographed, following post treatment care and attending all treatment and follow up visits.
4. The tattoo must include red pigment.

Exclusion Criteria:

1. Is female and pregnant, has been pregnant within the last 3 months, is currently breast feeding or planning a pregnancy during the study period.
2. Is hypersensitive to light exposure OR takes photo sensitized medication.
3. Has active or localized systemic infections.
4. Has a coagulation disorder or is currently using anti-coagulation medication (including but not limited to the heavy use of aspirin {greater than 81 mg per day}).
5. Has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
6. Is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within 3 months prior to entering this study.
7. Has used Accutane within 6 months prior to enrollment.
8. Has the need to be exposed to artificial tanning devices or excessive sunlight during the trial.
9. Has had prior treatment with parenteral gold therapy (gold sodium thiomalate).
10. Has a history of keloids.
11. Has evidence of compromised wound healing.
12. Has a history of basal cell carcinoma, squamous cell carcinoma or melanoma.
13. Has a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications or has an autoimmune disorder.
14. Is allergic to topical lidocaine or topical steroids.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Skin Care Physicians, Chestnut Hill, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Picosure Laser System
Started | 15
Completed | 8
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Picosure Laser System
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One of the subjects did not report his/her race/ethnicity.
  Participants
    Race/Ethnicity: number analyzed (Participants) | 14
    Race/Ethnicity: Caucasian | 10
    Race/Ethnicity: African American | 3
    Race/Ethnicity: Asian | 1
    Race/Ethnicity: Indian | 0
    Race/Ethnicity: Hispanic | 0
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is.
  The scale comes from this source:
  Gupta, Sharma. Skin typing: Fitzpatrick grading and others. Clinics in Dermatology. 2019;37(5):430-436. doi:10.1016/j.clindermatol.2019.07.010
  Participants
    Fitzpatrick Skin Type I | 2
    Fitzpatrick Skin Type II | 5
    Fitzpatrick Skin Type III | 4
    Fitzpatrick Skin Type IV | 0
    Fitzpatrick Skin Type V | 3
    Fitzpatrick Skin Type VI | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Tattoo Clearance
Description: Tattoo clearance will be measured using baseline and 2 month post treatment photos using a photographic scale. The scale ranges from 0 to 10, where 10 is 100% improvement from the baseline photo.
Time Frame: 2 months post last treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Picosure Laser System
Number analyzed (Participants) | 8
Participants
  # of Patients with 20% Improvement | 3
  # of Patients with 30% Improvement | 5

2. Secondary Outcome: Physician Satisfaction Questionnaire
Description: This measures the physician satisfaction from 1 to 5, where 5 is the most satisfied.
Time Frame: 2 months post last treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Picosure Laser System
Number analyzed (Participants) | 8
Participants
  Patients scored a 5 by physician | 4
  Patients scored a 4 by Physician | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the study duration, around 19 months.
Arm/Group | Picosure Laser System
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 15/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Picosure Laser System (N=15)
Pain (Nervous system disorders) | 8
Blistering (Skin and subcutaneous tissue disorders) | 7
Erythema (Skin and subcutaneous tissue disorders) | 5
Edema (Skin and subcutaneous tissue disorders) | 4
Bruising (Skin and subcutaneous tissue disorders) | 1
Pinpoint Bleeding (Skin and subcutaneous tissue disorders) | 4
Crusting (Skin and subcutaneous tissue disorders) | 11
Itching (Skin and subcutaneous tissue disorders) | 8
Allergic Reaction (Skin and subcutaneous tissue disorders) | 2
Hypopigmentation (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.